CLINICAL TRIAL: NCT05871346
Title: Effects of Complementary Feeding Counseling on Appropriate Complementary Feeding Practices and Child Undernutrition in West Gojjam Zone, Northwest Ethiopia: Cluster Randomized Controlled Trial
Brief Title: Effects of Complementary Feeding Counseling on Appropriate Complementary Feeding Practices and Child Undernutrition
Acronym: ACFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Shiferaw Birhanu Aynalem, MSc, Principal investigator., Bahir Dar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: adenek2195
Record Dates: First submitted 2023-04-07; First posted 2023-05-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Feeding Behavior
Keywords: Complementary feeding counseling (CFC); Appropriate complementary feeding practices (ACFP); Child Undernutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complementary Feeding Counseling (Experimental): Complementary feeding counseling to the mother-child pairs, in the intervention clusters, will be given by trained women development army (WDA) team leaders. The intervention process will have two components; training of WDA leaders, and counseling of mothers. Counselors' training will be given centrally by the principal investigator. During counseling, WDA leaders will use a counseling guide, which is prepared in Amharic, the local and the national language. The counseling guide contains seven key messages; complementary feeding: at 6 months, from 6-8 months, from 9-11 months, from 12-23 months, hygiene, breast feeding a sick child greater than 6 months, and signs that require mothers' special care of their children. Starting the children's 6 months of age, participants in the intervention group will receive in group counseling at convenient places, and individual counseling at each mother-child pair's home every month for 9 consecutive months (a total of 9 months follow up).
  Interventions: Behavioral: Complementary feeding counseling
- Routine Complementary Feeding Counseling (Experimental): Participants in the control clusters will receive the routine complementary feeding counseling, which is offered by heath extension workers and other health professionals.
  Interventions: Behavioral: Complementary feeding counseling

INTERVENTIONS:
Behavioral: Complementary feeding counseling — Complementary Feeding Counseling to Improve Appropriate Complementary Feeding Practices and Reduce Child Undernutrition

SUMMARY:
Appropriate complementary feeding practices as per the World Health Organization recommendations is a window of opportunity to promote health and prevent acute and chronic undernutrition (stunting, wasting & underweight). Globally, the burden of undernutrition remains unacceptably high, and the progress of undernutrition reduction is unsatisfactorily slow. In Ethiopia, appropriate complementary feeding practices of mothers to their children are very low. In contrast, child undernutrition is a major public health problem.

DETAILED DESCRIPTION:
Appropriate nutrition during the first 1000 days of life lays the foundation for a child's health and well-being. Introduction of complementary foods within 6-8 months of age and step-wise increase of diversified plant and animal-based diets is necessary, for which exclusive breast milk is no longer enough to meet the nutritional needs. Appropriate complementary feeding practices as per the World Health Organization recommendations is a window of opportunity to promote health and prevent acute and chronic undernutrition (stunting, wasting & underweight). Globally, the burden of undernutrition remains unacceptably high, and the progress of undernutrition reduction is unsatisfactorily slow. In Ethiopia, appropriate complementary feeding practices of mothers to their children are very low. In contrast, child undernutrition is a major public health problem. This study aims to determine the effects of complementary feeding counseling on appropriate complementary feeding practices and child undernutrition through a community-based randomized controlled trial.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Mother-child pairs whose children are 6 months old.
2. Mother-child pairs who reside in the study area for at least 6 months before the survey.
3. Mother-child pairs who have no intention of leaving the study area during the intervention period.

Exclusion Criteria:

1. Mothers with severe mental illness or who are unable to communicate (e.g., deaf).
2. Mother-child pairs with severe congenital malformations of their children.

Ages: 6 Months to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 776 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in appropriate complementary feeding practices of mothers for their children at 9 months. | Time Frame: At baseline (from June 9 to December 30, 2023), and in 9 months (from September 30 to December 30, 2024).
  Questions related to complementary feeding practices will be used to measure these practices of mothers for their children (Appropriate/Inappropriate). To measure appropriate complementary feeding practices, we will follow the World Health Organization recommendations for infant and young child feeding practices, continuation of breastfeeding, starting solid, semi-solid or soft foods at 6 months of age, the eight indicators used to calculate the dietary diversity, and the meal frequency will be asked. Minimum dietary diversity, minimum meal frequency, and consumption of egg and/or flesh food will be determined. Appropriate complementary feeding practice is defined if the four indicators: timely introduction of complementary foods, minimum dietary diversity, minimum meal frequency, and consumption of egg and/or flesh food are fulfilled. Otherwise, inappropriate if a child's feeding practices do not fulfill even one of the components of appropriate complementary feeding practices.

SECONDARY OUTCOMES:
Change from baseline in child nutritional status at 9 months | Time Frame: At baseline (from June 9 to December 30, 2023), and in 9 months (from September 30 to December 30, 2024).
  The child nutritional status (Undernutrition / No Undernutrition) will be determined by measuring the length, weight, and calculating the child's age. Length will be measured using a calibrated length board to the nearest 1mm (0.1cm). Weight will be measured using mechanical hanging scale with weighing pants to the nearest 10g at the time of enrollment and 100g at end-line measurements. Before weighing the child, the weighing scale will be hung securely and set to zero. The child's age will be calculated by subtracting the child's date of birth from the date of baseline data collection. Undernutrition will be defined if a child is considered wasted, or underweight, or stunted. The child is wasted: when the weight-for-length-Z score (WLZ) is <-2 standard deviations; underweight: when weight-for-age Z score (WAZ) is <-2 standard deviations, and stunted: when length-for-age Z score (LAZ) is <-2 standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Shiferaw Bi Aynalem, MSc, Principal Investigator — Bahir Dar University
Locations (1):
- Bahir Dar University, Bahir Dar, Amhara Regional State, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michaelsen KF, Grummer-Strawn L, Begin F. Emerging issues in complementary feeding: Global aspects. Matern Child Nutr. 2017 Oct;13 Suppl 2(Suppl 2):e12444. doi: 10.1111/mcn.12444. PMID 29032617